CLINICAL TRIAL: NCT02898948
Title: Procalcitonin (PCT) as a Diagnostic Marker of Bacterial Infection in the Patients Admitted for Fever and/or Inflammatory Syndrome to the Internal Medicine Department
Acronym: PCT-MI
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: RNI2015-38 Dr Schmidt
Record Dates: First submitted 2016-09-05; First posted 2016-09-13 (Estimated); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: Systemic Inflammatory Response Syndrome; Fever
Keywords: procalcitonin; bacterial infection
MeSH Terms: conditions — Systemic Inflammatory Response Syndrome; Fever; Bacterial Infections | interventions — Procalcitonin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Biological: Procalcitonin (PCT) as a diagnostic marker of bacterial infection

SUMMARY:
Levels of PCT (a marker of bacterial infection) are highest during sepsis: in fact, PCT is normally produced by the C cells in the thyroid gland. PCT was initially studied by Assicot1 for distinguishing between bacterial meningitis and viral meningitis. The CALC-I gene codes for PCT. In the absence of infection, the extrathyroid mRNA expression of the CALC-I gene is repressed, and expression is restricted to neuroendocrine thyroid and pulmonary cells. Infection induces the ubiquitous expression of the CALC-I gene. PCT is not transformed into calcitonin in parenchymatous tissues. In a context of sepsis, the whole body acts as a neuroendocrine gland. Sepsis upregulates PCT mRNA expression much more than that of other cytokines.

PCT is used in critical care departments as a diagnostic marker, a guide to treatment (antibiotics are withdrawn if the level falls) and a prognostic marker.

There are few data on the diagnostic use of PCT in an internal medicine department. The available studies yielded contradictory results and only one prospective study has been performed . The objective was to study PCT in non-infectious, inflammatory pathologies and to establish whether PCT could distinguish infections from other inflammatory pathologies in patients in an internal medicine department. In a ROC curve analysis, a PCT threshold of 0.35 µmol/l gave the greatest specificity (88%) and sensitivity (72%). Other studies have been performed but featured small sample sizes and a retrospective design.

Of the various studies performed in internal medicine departments, none included patients presenting with a suspected bacterial infection (according to the clinician's interpretation) and lacking information on their bacterial status. In fact, these diagnoses are a core component of hospitalisation in internal medicine departments for fever or inflammatory syndrome. The investigators intend to include all patients, including those lacking information on their microbiological status).

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 or over hospitalized in the internal medicine department at Amiens University Hospital, presenting with fever (>38.5°C) and/or inflammatory syndrome (CRP >5 mg/l) and having given their consent will be included.

Exclusion Criteria:

* Haemodialyzed patients.
* Age under 18.
* Legal guardianship.
* Refusal by the patient, or inability to give consent.
* Patients on antibiotics for more than 12 hours at the time of the PCT assay (the half-life of PCT is 22 hours, and the level falls rapidly when antibiotics are administered).
* PCT assays more than 12 hours after hospitalisation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 18 or over hospitalized in the internal medicine department at Amiens University Hospital, presenting with fever (>38.5°C) and/or inflammatory syndrome (CRP >5 mg/l)
Sampling Method: Non-Probability Sample
Enrollment: 116 (Actual)
Dates: Start 2016-02-11 (Actual); Primary Completion 2016-10-18 (Actual); Study Completion 2016-10-18 (Actual)

PRIMARY OUTCOMES:
PCT level | Day 0
  to determine whether PCT is a good diagnostic marker in patients presenting with fever and/or inflammatory syndrome

CONTACTS AND LOCATIONS:
Overall Officials: Jean SCHMIDT, MD, Principal Investigator — CHU Amiens
Locations (1):
- CHU Amiens, Amiens, France